CLINICAL TRIAL: NCT04134377
Title: High-Protein Food Snack and Albumin Outcomes in Hemodialysis Patients
Brief Title: High-Protein Food Snack for Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Fresenius Medical Care North America (Industry); National Kidney Foundation, United States (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201900310; AGR DTD 06-26-2019 (Other Grant/Funding Number: National Kidney Foundation); OCR21882 (Other: UF ID)
Record Dates: First submitted 2019-10-16; First posted 2019-10-22 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Renal Failure; Albumin; Double; Diet Habit
MeSH Terms: conditions — Renal Insufficiency; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Protein Food Snack (Experimental): Provide a high protein food snack the first 2 weeks of each month for 6 months. Each participant will receive an 8 ounce food snack after dialysis for a total of 6 food snacks for each month.
  Interventions: Other: Protein Food Snack

INTERVENTIONS:
Other: Protein Food Snack — The intervention is 6-months using a food snack with control being three months prior to and three months after-study invention whereby serum albumin levels will be collected monthly. If patients are participating in a supplement program, they will be maintained throughout all ten months of the study so long as the criteria for the supplement program (enrollment and discontinuation) is still being met.

SUMMARY:
The study team aims to provide a food snack that is high in protein (30 g) for two weeks each month (6 treatments per patient per month) for 6 consecutive months, post-dialysis treatment, to in-center hemodialysis patients of all vintages and with all levels and types of comorbidities. The study team will compare changes in serum albumin during the intervention (6 months) using the patients' own serum albumin results that are collected for three months prior to and three months after the intervention. Additionally, the study team will determine participants' dietary habits and appetite pre-, during and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Hemodialysis (CHD) therapy
* Active and permanent patients to the area Fresenius Kidney Care (FKC) Dialysis clinic
* No food allergies or dietary restrictions
* No contraindications to consuming anything by mouth as per the medical director and/or personal reporting.

Exclusion Criteria:

* Patients unable to commit to the full time commitments of the study
* Those who have food allergies, especially to Chicken, Pork Sausage, Eggs, Fresh Cilantro, Red and yellow bell peppers, Cucumbers, Mrs. Dash Grill Seasoning, Newman's Own Ranch Salad Dressing, Minced garlic, Sweet pickle relish, Vidalia onions, tomatoes
* Dietary restrictions as medically indicated,
* Trouble chewing/swallowing as confirmed by medical director, and/or personal reporting.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Serum albumin | Up to 12 months
  Change in grams of albumin per deciliter of blood (g/dL). Pre-, during, and 3-months post-intervention will complete monthly serum albumin lab draws.

SECONDARY OUTCOMES:
Serum phosphorus | Up to 12 months
  change in milligrams of phosphorus per deciliter of blood (mg/dL). Pre-, during, and 3-months post-intervention will complete monthly serum phosphorus lab draws.
Diet Intake | Up to 12 months
  This is a 9-item survey, "Diet Intake Survey", that obtains information about participants' appetites and dietary behaviors. Pre-, during, and 3-months post-intervention will complete monthly surveys on participants' diet habits to assess the impact the food snack has on total protein to calories.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette M Andrade, PhD, Principal Investigator — University of Florida
Locations (1):
- Fresenius Medical Care, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No